CLINICAL TRIAL: NCT04231851
Title: Phase II Study of the Combination of CPX-351 and Glasdegib in Previously Untreated Patients With Acute Myelogenous Leukemia With MDS Related Changes or Therapy-related Acute Myeloid Leukemia
Brief Title: CPX-351 and Glasdegib for Newly Diagnosed Acute Myelogenous Leukemia With MDS Related Changes or Therapy-related Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Jazz Pharmaceuticals (Industry); Pfizer (Industry)
Responsible Party: Principal Investigator, Deepa Jeyakumar, HS Associate Clinical Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20195533; UCI 18-105 (Other: UCI CFCCC); UCHMC1913 (Other: University of California Hematologic Malignancies Consortium)
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Acute Myelogenous Leukemia (AML) Due to Therapy; Acute Myeloid Leukemia With Myelodysplasia-Related Changes
Keywords: Therapy-Related AML; AML with MDS related changes
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — glasdegib; CPX-351; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CPX-351 and Glasdegib (Experimental): In Induction, subjects receive 44mg/m2/100mg/m2 IV on days 1, 3 and 5 and Glasdegib 100mg PO daily on days 6 to 28.
  If re-induction is needed: Subjects receive 44mg/m2/100mg/m2 IV on days 1 and 3 and Glasdegib 100mg PO daily on days 4 to 28.
  In consolidation: Subjects receive 29mg/m2/65mg/m2 IV on days 1 and 3 and Glasdegib 100mg PO daily on days 4 to 28.
  If maintenance is required, Subjects receive Glasdegib 100mg PO daily for up to one year
  Interventions: Drug: Glasdegib; Drug: CPX-351

INTERVENTIONS:
Drug: Glasdegib — Given PO
  Other Names: DAURISMO™
Drug: CPX-351 — Given IV
  Other Names: Daunorubicin and cytarabine; VYXEOS®

SUMMARY:
This is a phase 2 single-arm, open-label clinical trial determining efficacy of CPX-351 in combination with Glasdegib in subjects with Acute Myelogenous Leukemia with myelodysplastic syndrome related changes or therapy-related acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated therapy-related AML or AML with myelodysplastic related changes as described by World Health Organization (WHO) 2016

  1. AML arising in MDS (including CMML) or MDS/MPN syndrome
  2. AML with MDS-related cytogenetic abnormalities (Appendix A, metaphase FISH allowable as surrogate for cytogenetics)
  3. AML with multi-lineage dysplasia involving the presence of 50% or more dysplastic cells in at least two cell lines and in the absence of mutation in NPM1 or biallelic CEBPA (as per WHO 2016)
* Adults 18 years of age or older
* ECOG performance status 0 to 2
* Adequate organ function as defined as:

  1. Left Ventricular Ejection Fraction (LVEF) > 50%
  2. Serum total bilirubin < 2.0 mg/dL, unless considered due to Gilbert's disease or leukemic involvement
  3. AST, ALT and alkaline phosphatase < 3 times the upper limit of normal, unless considered due to leukemic involvement
  4. Serum creatinine < 2.0 mg/dL, or creatinine clearance > 40 mL/min based on Cockcroft-Gault GFR
* Absence of unstable cardiac disease defined as myocardial infarction within 6 months, uncontrolled heart failure, or uncontrolled cardiac arrhythmia
* Ability to understand and the willingness to sign a written informed consent or subject's legally authorize representative (LAR) has provided informed consent prior to any study-specific activities/procedures being initiated when the subject has any kind of condition that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication

  1. A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

     1. Has not undergone a hysterectomy or bilateral oophorectomy; or
     2. Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
  2. Women of child-bearing potential has negative pregnancy test within 72 hours of initiating study drug dosing
  3. Male subjects must agree to use a latex condom during sexual contact with females of childbearing potential even if they have had a successful vasectomy starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Leukapheresis, corticosteroid and hydroxyurea are permitted as initial management of hyperleukocytosis at the investigator's discretion for up to 7 days after starting study therapy. Hyperleukocytosis is defined as greater than 30k WBC. When possible, a bone marrow biopsy for screening should be performed prior to the initiation hyperleukocytosis

Exclusion Criteria:

* Prior treatment with Glasdegib or CPX-351
* Previously treated AML except for initial management of hyperleukocytosis. Treatment with hypomethylating therapy for MDS is allowable but not since their diagnosis of AML. No prior treatment with cytarabine or daunorubicin are allowed
* Concurrent FLT3 mutation that the treating physician deems necessary to treat with midostaurin, whereas patients with FLT3-mutated AML not treated with midostaurin can be enrolled. Patients with known Core Binding Factor -t(8;21), inv(16), t(16;16) are allowed for study participation at the treating investigator's discretion
* Active CNS or testicular involvement by leukemia; diagnostic lumbar puncture is not required
* History of neurologic disorder including but not limited to: prior seizure, epilepsy, structural brain abnormality, benign brain tumor, stroke, brain injuries, dementia, movement disorder or other significant CNS abnormalities
* Baseline QT corrected interval based on Fridericia's formula (QTcF) interval > 450 ms
* Acute coronary syndrome in the past 12 months, NYHA class III or VI
* Known history of Wilson's disease or other copper handling disorder
* History of GI malabsorptive disease
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Known HIV infection
* Active hepatitis B or hepatitis C infection (patients who successfully completed curative hepatitis C therapy can be enrolled)
* Any uncontrolled infection, active bacterial or viral infection manifesting as fevers or hemodynamic instability within the past 72 hours
* Proven active invasive fungal infection
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Severe or uncontrolled medical disorder that would, in the investigator's opinion, impair ability to receive study treatment (i.e., uncontrolled diabetes, chronic renal disease, chronic pulmonary disease or active, uncontrolled infection, psychiatric illness/social situations that would limit compliance with study requirements
* Current or anticipated use of other investigational agents
* For patients with prior anthracycline exposure, the cumulative life-time dose should not exceed 386mg/m2 at the time of study entry (to convert different anthracycline to daunorubicin-equivalent, see Appendix H for conversion factors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Event-Free Survival at 6 months | 6 months
  This is defined as the percentage of subjects with event-free survival (EFS) at 6 months. EFS is defined as the number of months where patients are in a remission state.

SECONDARY OUTCOMES:
Percentage of Grade 3-5 Adverse Events | From the start date of treatment until 4 weeks after removal of treatment due to disease progression, toxicity, delay of treatment, or withdrawal of treatment, whichever came first, an average of 1 year.
  To evaluate the tolerability of administering CPX-351 in combination with glasdegib in patients with newly diagnosed with Acute Myeloid Leukemia (AML) with Myelodysplastic Syndrome (MDS) related changes or treatment-related AML from the start of treatment, duration of treatment and up to 4 weeks after completion of study treatment. Toxicity and adverse events are based on the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0.
Overall Response Rate | From the start date of treatment until first date of CR/CRi or an average of 1 year.
  To assess the overall response rate to the combination of CPX-351 and glasdegib. The overall response rate (ORR) is defined as the rate of complete remissions (CR) and complete remission with incomplete count recovery (CRi). ORR = CR + CRi
Durability of Response | From the start date of treatment until first date of CR/CRi or an average of 1 year.
  Durability of response is measured by relapse-free survival (RFS). RFS is defined as the amount of time a patient remains in remission after having achieved a CR or CRi
Overall Survival of Patients who received the combination of CPX-351 and glasdegib | Time from screening biopsy for up to 12 months after the last patient is enrolled or until death from any cause, whichever came first.
  To evaluate the overall survival of patients with newly diagnosed with Acute Myeloid Leukemia (AML) with Myelodysplastic Syndrome (MDS) related changes or treatment-related AML.
Time to normal hematopoiesis as assessed by laboratory studies | From the start date of treatment until laboratory studies confirmation of normal hematopoiesis or an average of 1 year
  To evaluate the time to normal hematopoiesis, process by which blood cells are formed, as determined by laboratory studies inclusive of complete blood counts (CBCs)
Number of participants who go on to receive an allogenic hematopoietic stem cell transplant | Up to 3 years
  This is defined as the number of participants who continue on to receive an allogenic hematopoietic stem cell transplant after induction, re-induction, or consolidation.

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Jeyakumar, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (4):
- United States (4):
  - University of California, Los Angeles, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California